CLINICAL TRIAL: NCT05525780
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of Donepezil From Single Dose of GB-5001 Intramuscular Depot and Aricept® Oral Tablets (Pfizer Canada Inc.) in Healthy Male Volunteers
Brief Title: Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of Donepezil From Single Dose of GB-5001 IM Depot and Aricept® Oral Tablets in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: G2GBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G2GBio
Record Dates: First submitted 2022-08-23; First posted 2022-09-02 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Cohort Studies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GB-5001 (Experimental): GB-5001 Suspension for intramuscular (IM) injection at three doses
  Interventions: Drug: GB-5001
- Placebo (Placebo Comparator): Placebo Suspension for intramuscular (IM) injection, Volume to be matched with the active drug in the respective cohort
  Interventions: Drug: Placebo
- Oral cohort (Active Comparator): Aricept® tablet
  Interventions: Drug: Oral cohort

INTERVENTIONS:
Drug: GB-5001 — Depending on the cohort, volume will be varied to administer.
  Arms: GB-5001
Drug: Placebo — A matched volume of placebo product will be administered to each subject in each cohort.
  Arms: Placebo
Drug: Oral cohort — Single dose of Aricept tablet
  Arms: Oral cohort

SUMMARY:
This study is to evaluate the safety and tolerability of single dose of GB-5001 (donepezil) IM depot in healthy male volunteers. And, it is to predict the multiple-dose pharmacokinetics based on the single-dose pharmacokinetics of GB-5001 IM depot and the oral Aricept® (donepezil hydrochloride) tablet by PK modeling.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male volunteers, 18-55 years of age, inclusive at the time of informed consent.
* Body mass index (BMI) that is within 18.5 - 30.0 kg/m2, inclusive, and weight at least 55 kg and above.
* Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
* Systolic blood pressure between 95-140 mmHg, inclusive, and diastolic blood pressure between 55-90 mmHg, inclusive, and heart rate between 60-100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
* Clinical laboratory values within the clinical site's most recent acceptable laboratory test range, and/or values are deemed by the PI/Sub-Investigator as "Not Clinically Significant".

Exclusion Criteria:

* Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
* Known history or presence of seizure or convulsion, unless determined as not clinically significant by the PI/Sub-Investigator.
* Known history or presence of peptic ulcer or gastrointestinal bleeding within 3 months prior to study drug administration, unless determined as not clinically significant by the PI/Sub-Investigator.
* Known risk of developing ulcers (for example, if you are taking non-steroidal anti-inflammatory drugs [NSAIDS] or high doses of acetylsalicylic acid [ASA] [Aspirin®]), unless determined as not clinically significant by the PI/Sub-Investigator.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug experienced within 7 days prior to study drug administration, as determined by the PI/Sub-Investigator.
* Presence of any clinically significant illness within 30 days prior to dosing, as determined by the PI/Sub-Investigator
* Presence of any clinically significant illness within 30 days prior to dosing, as determined by the PI/Sub-Investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and dose-relationship of AEs | Day 64
Vital signs | Day 64
  blood pressure [BP], respiratory rate [RR], heart rate [HR], and temperature
Electrocardiograms | Day 64
Physical examination | Day 64
  Height, weight, and BMI will be recorded
Injection site assessments | Day 64

SECONDARY OUTCOMES:
Key PK parameters for single dose IM and Oral cohorts | Day 64
  AUCt: area under the plasma concentration vs time curve from time 0 to the time of the last measurable concentration
Key PK parameters for single dose IM and Oral cohorts | Day 64
  Cmax: maximum observed plasma concentration
Key PK parameters for single dose IM and Oral cohorts | Day 64
  tmax: time to maximum observed plasma concentration
Key PK parameters for single dose IM and Oral cohorts | Day 64
  λz: terminal elimination rate constant
Key PK parameters for single dose IM and Oral cohorts | Day 64
  t½: terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Québec, Canada

REFERENCES:
- [Derived] Khwarg J, Lee H, Yu KS, Seol E, Chung JY. Population Pharmacokinetic Modeling and Simulation for Dose Optimization of GB-5001, a Long-Acting Intramuscular Injection of Donepezil, in Healthy Participants. Neurol Ther. 2024 Oct;13(5):1453-1466. doi: 10.1007/s40120-024-00643-4. Epub 2024 Aug 10. PMID 39126603